CLINICAL TRIAL: NCT00868738
Title: Evaluation of Calcium, Vitamin D, Magnesium, and Zinc Absorption in Healthy Children 4 to 8 Years of Age
Brief Title: Evaluation of Calcium, Vitamin D, Magnesium, and Zinc Absorption in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Steve Abrams, Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: H-24134; 6250-51000-045-00D
Record Dates: First submitted 2009-03-24; First posted 2009-03-25 (Estimated); Last update posted 2011-11-02 (Estimated); Status verified 2011-11

CONDITIONS: Mineral Absorption
Keywords: Calcium; Vitamin D; Magnesium; Zinc
MeSH Terms: interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D (Active Comparator): Subjects will be provided supplemental vitamin D3 (1000 IU), given once daily as a softgel or liquid. Subjects will be instructed to take the supplement daily for 8 weeks.
  Interventions: Dietary Supplement: Vitamin D
- Placebo (Placebo Comparator): Subjects will be provided a placebo, given once daily as a softgel or liquid. Subjects will be instructed to take the supplement daily for 8 weeks.
  Interventions: Dietary Supplement: Vitamin D

INTERVENTIONS:
Dietary Supplement: Vitamin D — Subjects will be provided supplemental vitamin D3 (1000 IU) or placebo, given once daily (based on the stratification noted above). Vitamin D/placebo will be provided using a softgel or liquid. Subjects will be instructed to take the supplement daily for 8 weeks.

SUMMARY:
The goal of our research is to provide data to enhance the development of nutritional guidelines, especially as related to mineral nutrition, in children. Using human experimentation, we are studying methods of delivering the key minerals of calcium, zinc and iron in the diet so as to optimize health outcomes. We will conduct a controlled trial of vitamin D supplementation to assess the effects of vitamin D status on calcium absorption in small children. We will evaluate the effects of differing intakes of zinc on zinc and copper absorption. These studies will utilize stable isotope techniques so as to provide accurate, practically applicable information which may be obtained from the study populations in a safe manner. These data will have global application and provide a strong basis for evidence-based nutritional recommendations to be developed.

Objective #1: To evaluate the effects of supplemental vitamin D in enhancing calcium absorption in healthy children 4 to 8 yrs of age.

Objective #2: Assess the absorption of magnesium and zinc in healthy children 4 to 8 yrs of age.

DETAILED DESCRIPTION:
We plan to stratify subjects for randomization to either vitamin D supplements or placebo by serum 25-hydroxyvitamin D (25 OHD) into three groups: 0-20 ng/mL, 20-32 ng/mL, and >32 ng/mL.

There is no group assignment or randomization for the magnesium and zinc aspects of the study.

SCREENING VISIT: At the time of enrollment, subjects and their families will be asked to come to the General Clinical Research Center (GCRC) of Texas Children's Hospital for a screening visit. Prior to this visit, demographics from the parent/guardian will be recorded including the child's approximate height and weight, and the study dietitian will obtain two 24-hour dietary recalls from the parent to determine calcium intake for enrollment. During this screening visit, informed written consent will be obtained, a medical history taken, and a physical examination performed.

The study dietitian will instruct the parent/guardian and child on the use of a food scale to weigh and record dietary intake for a 3-day period (ie, 3-day weighed diet record). The 3-day weighed diet record will begin the following day. This method has been shown to provide the best estimate of dietary intakes in children (Crawford PB et al, J Am Diet Assoc. 1994; 94:626-630; Fisher JO et al, Am J Clin Nutr. 2008; 88:407-415). Upon analysis of their child's intake, parents will be instructed to maintain a similar nutrient intake throughout the study. Compliance will be monitored via 3-day weighed home diet records timed with their other study visits. If analysis shows that the child's intake has significantly changed (± 20% of a nutrient), the parent will be counseled by the study dietitian on readjusting the child's intake back to the usual level determined at baseline.

In addition, the study dietitian will prepare sample menus based on the child's food preferences and dietary intake levels and provide them to the parent. Parents can use the sample menus to assist them in maintaining the child's usual mineral intake.

STUDY VISIT 1: Subjects and a parent/guardian will return to the GCRC for a 24-hour overnight stay, arriving in the morning for a baseline stable isotope study. We will utilize the dual-tracer stable isotope technique as in our previous studies. At this visit subjects will receive intravenous isotope doses 1 mg 42Ca, 6 mg 25Mg, and 0.4 mg 70Zn. At the time of the IV isotope, we will collect a blood sample (10mL for serum calcium, phosphorus, alkaline phosphatase, magnesium, 25OHD, 1,25-dihydroxyvitamin D, hepcidin, ferritin, TIBC, transferrin saturation, hemoglobin, hematocrit, and RBC indices). Topical numbing cream or spray to minimize pain at the injection site will be offered to all subjects.

A dual-energy x-ray absorptiometry (DEXA) measurement of total body bone mineral content/density and body fat will be made. This is done to use as a covariate in evaluating vitamin D levels and calcium absorption.

A 24-hr urine collection while they stay inpatient will begin with the timing of the first isotope. After they are discharged, subjects will be instructed on collecting another 48-hr urine collection (72-hr total) at home as well as a final spot urine at 96 hours after the first isotope.

Subjects will receive oral isotopes (20 mcg 46Ca, 12 mg 26Mg, and 2 mg 67Zn) mixed with 120 mL of calcium and vitamin D-fortified orange juice or milk. The breakfast will be a fixed meal providing a total of ~300 mg calcium. Lunch will provide ~300mg calcium; dinner will provide ~300mg calcium (totaling ~900mg calcium). All meals at the GCRC will be pre- and post-weighed to determine actual intake. After discharge, subjects will record dietary intake using another 3-day weighed diet record.

Approximately one week after Study Visit 1, the results from the serum 25OHD test will be back and we will stratify subjects accordingly into three groups: 0-20 ng/mL, 20-32 ng/mL, and >32 ng/mL. Subjects will return to the CNRC to be provided supplemental vitamin D3 (1000 IU) or placebo, given once daily (based on the stratification noted above). Vitamin D/placebo will be provided using a softgel or liquid. Subjects will be instructed to take the supplement daily for 8 weeks. They will be provided with study calendars to mark daily when they remember to take the supplement. Calendars and remaining supplements will be returned to the study center for counting to determine compliance.

Subjects will return urine samples, food scales, and diet records to the study personnel at the CNRC. The CNRC driver may also be utilized for the purpose of picking up samples or delivering the supplement. Periodic phone calls will be made to the home of the subject to monitor compliance with taking the supplement.

STUDY VISIT 2: Eight (8) weeks after the subjects began taking their supplement, subjects will return to the GCRC for a repeat study of absorption. Prior to this visit, subjects will receive a food scale and will perform another 3-day weighed diet record to demonstrate consistency of diet throughout the study period. Subjects will again arrive in the morning to the GCRC for a 24-hr inpatient study visit. They will bring with them all study calendars and remaining supplements for compliance monitoring. Study Visit 2 is similar in all aspects of Study Visit 1 regarding the calcium and vitamin D portion of the study. Magnesium and zinc measurements will not be repeated at Study Visit 2.

At this visit subjects will receive an intravenous isotope dose of 1 mg 42Ca. At the time of the IV isotope, we will collect a blood sample (same labs as in Study Visit 1). Topical numbing cream or spray to minimize pain at the injection site will be offered to all subjects.

A 24-hr urine collection while they stay inpatient will begin with the timing of the first isotope. After they are discharged, subjects will not be required to continue any additional urine collections.

Subjects will receive 20 mcg 46Ca stable isotope mixed with 120 mL of calcium and vitamin D-fortified orange juice or milk. The breakfast will be a fixed meal providing a total of ~300 mg calcium. Lunch will provide ~300mg calcium; dinner will provide ~300mg calcium (totaling ~900mg calcium). All meals at the GCRC will be pre- and post-weighed to determine actual intake.

Upon discharge, subjects will discontinue the supplementation and the study will be complete.

In interpreting the results, we will note ethnicity, the season of measurement and qualitative descriptions of sun exposure by considering the amount of time spent outside. However, we will not specifically assess sun exposure as this is not practical in small children. In general, we would not expect large changes in these in Houston during the 8 weeks of the study, but will ensure that the two studies do not cross a period of major change such as having the first study done before summer camp and the second right afterwards.

Urine and serum samples will be prepared for mass spectrometric analysis using an oxalate precipitation technique. Samples will be analyzed for isotopic enrichment using a magnetic sector ICP-MS. This is a high-speed instrument capable of analysis of the desired ratio with precision and accuracy of 0.3-0.5%.

Contingencies: We do not anticipate any problems with this study that would require changing or altering the protocol. Our sample size does not allow us to evaluate gender or ethnicity separately to determine differences in effects among these. There is no reason to expect differences in vitamin D effects on calcium absorption based on these (Weaver, personal communication). Additionally, dietary recommendations reflect the diversity of our population and if we identify trends towards specific ethnic or gender effects we can study this further in future population studies. This study will look at absorption only as an endpoint. If a benefit is found, we will develop a long-term trial evaluating bone mineral outcomes. However, this would require larger groups and a full year of study and is beyond the scope of this initial study. If no difference in calcium absorption is shown with 1000 IU/d of vitamin D, it is extremely unlikely that an effect on bone mineral would be found justifying a long-term study.

Magnesium absorption studies require a full 72-hour urine collection for accuracy. It is not practical to keep children this age in-patient for this time so after 24 hours, collections will be done at home. We have extensive experience with assisting families in home urine collections. There is the possibility of some loss of urine in a 72-hour collection. However, in that case we would continue the collection as the method's accuracy is not highly sensitive to the loss of a single or a small number of urine specimens in small children. Magnesium balance is not regulated by endogenous excretion (similar to calcium) and thus the absorption studies will provide adequate information to estimate net balance.

Subjects may be told their weight and height measurements at each visit to the GCRC. All other study related information will be held until the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Delivery at > or = 35.0 weeks gestation with birth weight > or = 2.5 kg
* BMI: 10th - 90th percentile for age and gender
* Ages 4.0 to 8.9 years
* Ethnic distribution of greater Houston area
* Usual calcium intake 600-1200 mg/d based on two 24-hour dietary recalls by phone
* Any regularly taken (daily) vitamins and minerals must be stopped at least 1 month before starting the study

Exclusion Criteria:

* History of any chronic illness.
* Regularly taken (daily) medications (except seasonal allergies).
* Avoidance of dairy products or meat in the diet.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2009-03; Primary Completion 2011-08 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
To evaluate the effects of supplemental vitamin D in enhancing calcium absorption in healthy children 4 to 8 yrs of age. | End of the study

SECONDARY OUTCOMES:
Assess the absorption of magnesium and zinc in healthy children 4 to 8 yrs of age. | End of the study

CONTACTS AND LOCATIONS:
Overall Officials: Steve Abrams, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine / Texas Children's Hospital, Houston, Texas, United States

REFERENCES:
- [Background] Abrams SA, Griffin IJ, Hawthorne KM, Liang L, Gunn SK, Darlington G, Ellis KJ. A combination of prebiotic short- and long-chain inulin-type fructans enhances calcium absorption and bone mineralization in young adolescents. Am J Clin Nutr. 2005 Aug;82(2):471-6. doi: 10.1093/ajcn.82.2.471. PMID 16087995
- [Background] Abrams SA, Hawthorne KM, Aliu O, Hicks PD, Chen Z, Griffin IJ. An inulin-type fructan enhances calcium absorption primarily via an effect on colonic absorption in humans. J Nutr. 2007 Oct;137(10):2208-12. doi: 10.1093/jn/137.10.2208. PMID 17884999
- [Background] Ames SK, Gorham BM, Abrams SA. Effects of high compared with low calcium intake on calcium absorption and incorporation of iron by red blood cells in small children. Am J Clin Nutr. 1999 Jul;70(1):44-8. doi: 10.1093/ajcn/70.1.44. PMID 10393137
- [Background] Beard JL, Dawson H, Pinero DJ. Iron metabolism: a comprehensive review. Nutr Rev. 1996 Oct;54(10):295-317. doi: 10.1111/j.1753-4887.1996.tb03794.x. PMID 9063021
- [Background] Bischoff-Ferrari HA, Dietrich T, Orav EJ, Dawson-Hughes B. Positive association between 25-hydroxy vitamin D levels and bone mineral density: a population-based study of younger and older adults. Am J Med. 2004 May 1;116(9):634-9. doi: 10.1016/j.amjmed.2003.12.029. No abstract available. PMID 15093761
- [Background] Bray MS, Shaw CA, Moore MW, Garcia RA, Zanquetta MM, Durgan DJ, Jeong WJ, Tsai JY, Bugger H, Zhang D, Rohrwasser A, Rennison JH, Dyck JR, Litwin SE, Hardin PE, Chow CW, Chandler MP, Abel ED, Young ME. Disruption of the circadian clock within the cardiomyocyte influences myocardial contractile function, metabolism, and gene expression. Am J Physiol Heart Circ Physiol. 2008 Feb;294(2):H1036-47. doi: 10.1152/ajpheart.01291.2007. Epub 2007 Dec 21. PMID 18156197
- [Background] Davidsson L, Ziegler EE, Kastenmayer P, Hurrell RF. Erythrocyte incorporation of iron by infants: iron bioavailability from a low-iron infant formula and an evaluation of the usefulness of correcting erythrocyte incorporation values, using a reference dose or plasma ferritin concentrations. Br J Nutr. 2000 Dec;84(6):847-53. PMID 11177201
- [Background] Donovan A, Andrews NC. The molecular regulation of iron metabolism. Hematol J. 2004;5(5):373-80. doi: 10.1038/sj.thj.6200540. PMID 15448662
- [Background] Eisenstein RS. Iron regulatory proteins and the molecular control of mammalian iron metabolism. Annu Rev Nutr. 2000;20:627-62. doi: 10.1146/annurev.nutr.20.1.627. PMID 10940348
- [Background] Fleet JC, Eksir F, Hance KW, Wood RJ. Vitamin D-inducible calcium transport and gene expression in three Caco-2 cell lines. Am J Physiol Gastrointest Liver Physiol. 2002 Sep;283(3):G618-25. doi: 10.1152/ajpgi.00269.2001. PMID 12181175
- [Background] Fleet JC, Wood RJ. Specific 1,25(OH)2D3-mediated regulation of transcellular calcium transport in Caco-2 cells. Am J Physiol. 1999 Apr;276(4):G958-64. doi: 10.1152/ajpgi.1999.276.4.G958. PMID 10198340
- [Background] Friend DR. Drug delivery to the small intestine. Curr Gastroenterol Rep. 2004 Oct;6(5):371-6. doi: 10.1007/s11894-004-0052-z. PMID 15341712
- [Background] Garcia-Casal MN, Leets I, Layrisse M. Beta-carotene and inhibitors of iron absorption modify iron uptake by Caco-2 cells. J Nutr. 2000 Jan;130(1):5-9. doi: 10.1093/jn/130.1.5. PMID 10613757
- [Background] Gordon CM, DePeter KC, Feldman HA, Grace E, Emans SJ. Prevalence of vitamin D deficiency among healthy adolescents. Arch Pediatr Adolesc Med. 2004 Jun;158(6):531-7. doi: 10.1001/archpedi.158.6.531. PMID 15184215
- [Background] Griffin IJ, Davila PM, Abrams SA. Non-digestible oligosaccharides and calcium absorption in girls with adequate calcium intakes. Br J Nutr. 2002 May;87 Suppl 2:S187-91. doi: 10.1079/BJNBJN/2002536. PMID 12088517
- [Background] Griffin IJ, Lynch MF, Hawthorne KM, Chen Z, Hamzo M, Abrams SA. Magnesium retention in 12 to 48 month-old children. J Am Coll Nutr. 2008 Apr;27(2):349-55. doi: 10.1080/07315724.2008.10719711. PMID 18689570
- [Background] Griffin IJ, Lynch MF, Hawthorne KM, Chen Z, Hamzo MG, Abrams SA. Zinc homeostasis in 1-4 year olds consuming diets typical of US children. Br J Nutr. 2007 Aug;98(2):358-63. doi: 10.1017/S0007114507708796. Epub 2007 Apr 26. PMID 17459190
- [Background] Gunshin H, Allerson CR, Polycarpou-Schwarz M, Rofts A, Rogers JT, Kishi F, Hentze MW, Rouault TA, Andrews NC, Hediger MA. Iron-dependent regulation of the divalent metal ion transporter. FEBS Lett. 2001 Dec 7;509(2):309-16. doi: 10.1016/s0014-5793(01)03189-1. PMID 11741608
- [Background] Hallberg L, Rossander L, Skanberg AB. Phytates and the inhibitory effect of bran on iron absorption in man. Am J Clin Nutr. 1987 May;45(5):988-96. doi: 10.1093/ajcn/45.5.988. PMID 3034044
- [Background] Heaney RP, Dowell MS, Hale CA, Bendich A. Calcium absorption varies within the reference range for serum 25-hydroxyvitamin D. J Am Coll Nutr. 2003 Apr;22(2):142-6. doi: 10.1080/07315724.2003.10719287. PMID 12672710
- [Background] Holick MF. Sunlight and vitamin D for bone health and prevention of autoimmune diseases, cancers, and cardiovascular disease. Am J Clin Nutr. 2004 Dec;80(6 Suppl):1678S-88S. doi: 10.1093/ajcn/80.6.1678S. PMID 15585788
- [Background] Johnston CC Jr, Miller JZ, Slemenda CW, Reister TK, Hui S, Christian JC, Peacock M. Calcium supplementation and increases in bone mineral density in children. N Engl J Med. 1992 Jul 9;327(2):82-7. doi: 10.1056/NEJM199207093270204. PMID 1603140
- [Background] Lynch MF, Griffin IJ, Hawthorne KM, Chen Z, Hamzo M, Abrams SA. Calcium balance in 1-4-y-old children. Am J Clin Nutr. 2007 Mar;85(3):750-4. doi: 10.1093/ajcn/85.3.750. PMID 17344496
- [Background] Lynch SR. Iron overload: prevalence and impact on health. Nutr Rev. 1995 Sep;53(9):255-60. doi: 10.1111/j.1753-4887.1995.tb05482.x. PMID 8577408
- [Background] McKie AT, Barrow D, Latunde-Dada GO, Rolfs A, Sager G, Mudaly E, Mudaly M, Richardson C, Barlow D, Bomford A, Peters TJ, Raja KB, Shirali S, Hediger MA, Farzaneh F, Simpson RJ. An iron-regulated ferric reductase associated with the absorption of dietary iron. Science. 2001 Mar 2;291(5509):1755-9. doi: 10.1126/science.1057206. Epub 2001 Feb 1. PMID 11230685
- [Background] Monsen ER. Iron nutrition and absorption: dietary factors which impact iron bioavailability. J Am Diet Assoc. 1988 Jul;88(7):786-90. PMID 3290310
- [Background] Northstone K, Emmett P. Multivariate analysis of diet in children at four and seven years of age and associations with socio-demographic characteristics. Eur J Clin Nutr. 2005 Jun;59(6):751-60. doi: 10.1038/sj.ejcn.1602136. PMID 15841093
- [Background] Rajakumar K, Fernstrom JD, Holick MF, Janosky JE, Greenspan SL. Vitamin D status and response to Vitamin D(3) in obese vs. non-obese African American children. Obesity (Silver Spring). 2008 Jan;16(1):90-5. doi: 10.1038/oby.2007.23. PMID 18223618
- [Background] Thane CW, Bates CJ, Prentice A. Risk factors for low iron intake and poor iron status in a national sample of British young people aged 4-18 years. Public Health Nutr. 2003 Aug;6(5):485-96. doi: 10.1079/PHN2002455. PMID 12943565
- [Background] Vieth R, Bischoff-Ferrari H, Boucher BJ, Dawson-Hughes B, Garland CF, Heaney RP, Holick MF, Hollis BW, Lamberg-Allardt C, McGrath JJ, Norman AW, Scragg R, Whiting SJ, Willett WC, Zittermann A. The urgent need to recommend an intake of vitamin D that is effective. Am J Clin Nutr. 2007 Mar;85(3):649-50. doi: 10.1093/ajcn/85.3.649. No abstract available. PMID 17344484
- [Background] Walczyk T, Davidsson L, Rossander-Hulthen L, Hallberg L, Hurrell RF. No enhancing effect of vitamin A on iron absorption in humans. Am J Clin Nutr. 2003 Jan;77(1):144-9. doi: 10.1093/ajcn/77.1.144. PMID 12499334
- [Background] Wessling-Resnick M. Iron transport. Annu Rev Nutr. 2000;20:129-51. doi: 10.1146/annurev.nutr.20.1.129. PMID 10940329
- [Background] Zoller H, Theurl I, Koch R, Kaser A, Weiss G. Mechanisms of iron mediated regulation of the duodenal iron transporters divalent metal transporter 1 and ferroportin 1. Blood Cells Mol Dis. 2002 Nov-Dec;29(3):488-97. doi: 10.1006/bcmd.2002.0587. PMID 12547239
- [Derived] Huey SL, Acharya N, Silver A, Sheni R, Yu EA, Pena-Rosas JP, Mehta S. Effects of oral vitamin D supplementation on linear growth and other health outcomes among children under five years of age. Cochrane Database Syst Rev. 2020 Dec 8;12(12):CD012875. doi: 10.1002/14651858.CD012875.pub2. PMID 33305842
- [Derived] Cummings SR, Eastell R. A History of Pivotal Advances in Clinical Research into Bone and Mineral Diseases. J Bone Miner Res. 2018 Jan;33(1):5-12. doi: 10.1002/jbmr.3353. Epub 2018 Jan 12. No abstract available. PMID 29329487
- [Derived] Abrams SA, Hawthorne KM, Chen Z. Supplementation with 1000 IU vitamin D/d leads to parathyroid hormone suppression, but not increased fractional calcium absorption, in 4-8-y-old children: a double-blind randomized controlled trial. Am J Clin Nutr. 2013 Jan;97(1):217-23. doi: 10.3945/ajcn.112.046102. Epub 2012 Nov 14. PMID 23151536